CLINICAL TRIAL: NCT02662725
Title: A Multicenter Phase II Study of Ipilimumab Combined With a Stereotactic Radiosurgery in Melanoma Patients With Brain Metastases
Brief Title: Ipilimumab Combined With a Stereotactic Radiosurgery in Melanoma Patients With Brain Metastases
Acronym: IPI+RTS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011_48; 2012-000852-32 (EudraCT Number)
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Melanoma; Brain Metastasis
Keywords: melanoma; brain metastasis; stereotactic radiosurgery; Ipilimumab; survival; safety; efficacy
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — Ipilimumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ipilimumab + Stereotactic Radiosurgery (Experimental): ipilimumab combined with a Stereotactic Radiosurgery in Melanoma Patients with Brain Metastases
  Interventions: Drug: IPILIMUMAB; Radiation: Stereotactic radiosurgery

INTERVENTIONS:
Drug: IPILIMUMAB
Radiation: Stereotactic radiosurgery

SUMMARY:
This is a non-controlled, open label, Phase II Study of ipilimumab combined with a Stereotactic Radiosurgery. The study included an induction phase of four IV infusions of Ipilimumab at 10 mg/kg every 3 weeks associated with a stereotactic radiosurgery performed 3 days before 2nd ipilimumab administration. A Maintenance phase included Ipilimumab, IV, 10 mg/kg once every 12 weeks, starting at week 24, in the absence of PD, unacceptable toxicity or withdrawal of consent or disease progression. The primary objective is the overall survival. The Secondary objectives include safety, ORR, PFS and peripheral blood absolute lymphocyte count (ALC) as a predictive biomarker.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent.
2. Men and women ≥ 18 years of age.
3. Patient eligible to single dose Stereotactic Radiotherapy (Radiosurgery) as per the pluridisciplinary committee.
4. Neurologically asymptomatic or pauci-symptomatic patients. Patients with moderated neurological symptoms without systemic corticosteroids treatment can be included.
5. Less than 4 brain metastasis at the MRI. Brain metastasis should measure less than 3 cm in diameter. At least one brain metastasis > 5mm.
6. Maximum one prior systemic therapy for metastatic disease is allowed.
7. Prior treatment with INTERFERON in the adjuvant setting is authorized. Prior treatment with anti-CTLA-4 is NOT authorized.
8. ECOG Performance Status 0 or 1
9. Within the last 2 weeks prior to study day 1 the following laboratory parameters, which should be within the ranges specified:

Exclusion Criteria:

1. The patient requires concomitant chronic treatment with systemic corticosteroids or any other immunosuppressive agents 7 days prior to inclusion.
2. Neurological symptoms treated with systemic corticosteroids (whatever the dose of corticoids).
3. The patient has concurrent severe medical problems, unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk such as but not limited to: Cardiac insufficiency (III or IV as per NYHA classification), Renal insufficiency, ongoing infection.
4. Any symptom of concomitant tumour meningitis
5. History of immediate or delayed gadolinium hypersensitivity, or any contraindication to undergo MRI examination (Pacemaker, brain aneurysms clips)
6. Any concurrent malignancy other than non-melanoma skin cancer, or carcinoma in situ of the cervix (Subjects with a previous malignancy but without evidence of disease for 5 years will be allowed to enter the study)
7. Uncontrolled infectious diseases - requires negative tests for clinically suspected HIV, HBV and HCV. If positive results are not indicative of true active or chronic infection, the subject may enter the study after discussion and agreement between the Investigator and the Medical Monitor.
8. Active autoimmune disease. Autoimmune disease: subjects with a documented history of inflammatory bowel disease, including ulcerative colitis and Crohn's disease are excluded from this study as are subjects with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], Systemic Lupus Erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]).
9. Subjects with motor neuropathy considered of autoimmune origin (e.g., Guillain Barré Syndrome) are excluded from this study
10. Previous treatment with a CTLA-4 antagonist agent, including treatment in adjuvant setting.
11. The patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent or to comply with the trial procedures.
12. Lack of availability for clinical follow-up assessments.
13. For female patients: the patient is pregnant or lactating.
14. Women of childbearing potential: refusal or inability to use effective means of contraception
15. Participation in another clinical trial protocol within 30 days prior to enrolment
16. Persons protected by a legal regime (guardianship, trusteeship)
17. Patients in emergency situations
18. Patients kept in detention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2012-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Overall survival rate | until week 96 or death

SECONDARY OUTCOMES:
All adverse events ≥ Grade 3 according to CTCAE, Version 4.0 criteria, | through study completion, until week 96
Overall response rate in brain | until week 96 or death
  according to immune-related response criteria (ir-RC) and the mWHO criteria of target lesion
Global overall response rate | until week 96 or death
  according to immune-related response criteria (ir-RC) and the mWHO criteria of target lesions
Disease control rate in brain | until week 96 or death
  according to immune-related response criteria (ir-RC) and the mWHO criteria of target lesions
Global disease control rate | until week 96 or death
  according to immune-related response criteria (ir-RC) and the mWHO criteria of target lesions
Progression free survival | until week 96 or death

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Mortier, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (18):
- France (18):
  - CHU de Bordeaux, Bordeaux
  - CHU de Caen, Caen
  - Hôpital Trousseau - CHRU de Tours, Chambray-lès-Tours
  - CHU - Hôpital d'Estaing, Clermont-Ferrand
  - Hôpital A. Michallon, La Tronche
  - CHRU, Hôpital Claude Huriez, Lille
  - AP-HM Hôpital de la Timone, Marseille
  - Hôpital Saint Eloi, Montpellier
  - CHU Nantes - Place Alexis Ricordeau, Nantes
  - Hôpital Archet 2, Nice
  - AP-HP, Hôpital Ambroise Paré, Paris
  - AP-HP, Hôpital Saint-Louis, Paris
  - CHU de Bordeaux, Pessac
  - Centre hospitalier Lyon Sud, Pierre-Bénite
  - Centre Régional de Lutte Contre le Cancer Eugène Marquis, Rennes
  - CHU de Toulouse - Larrey, Toulouse
  - Hôpitaux de Brabois, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No